CLINICAL TRIAL: NCT05929625
Title: Radiofrequency and Ultrasound for Improvement of Skin Laxity and Wrinkles: Efficacy and Safety Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BTL-585F_100
Record Dates: First submitted 2023-04-11; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Intervention Model Description: The study is a prospective multicenter single-blinded two-arm study. The subjects will be enrolled and assigned into two study groups; group A (RF & US) and B (only RF) which will receive a treatment with different settings.
Who Masked: Participant
Masking Description: The study design is single blinded; only the subject will be unaware of the group assignment. The operator providing the treatment will be aware of the subject's group assignment and will perform the treatment with the setting according to the subject's group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- RF+US group (Experimental): Subjects will be treated with the subject device using both, radiofrequency and ultrasound energies simultaneously with regular treatment settings.
  Interventions: Device: BTL-585-2 RF+US
- RF only group (Experimental): Subjects will be treated with the subject device using only radiofrequency energy with regular treatment settings.
  Interventions: Device: BTL-585-2 RF

INTERVENTIONS:
Device: BTL-585-2 RF+US — The subjects of RF+US group will receive four simultaneous RF+US treatments of the entire face area including forehead, upper and lower cheeks and area around eyes.
  Arms: RF+US group
Device: BTL-585-2 RF — The subjects of RF only study group will receive four RF treatments of the entire face area including forehead, upper and lower cheeks and area around eyes.
  Arms: RF only group

SUMMARY:
This study will evaluate the clinical efficacy, safety and the performance of radiofrequency heating and ultrasound delivered by the BTL-585-2 applicator of the BTL-585F system for non-invasive treatment of facial wrinkles and correcting facial skin laxity. The study is a prospective multicenter single-blinded two-arm study. The subjects will be enrolled and assigned into two study groups; group A (RF & US) and B (only RF) which will receive a treatment with different settings. Subjects of both groups will be required to complete four (4) treatment visits and two to three follow-up visits.

DETAILED DESCRIPTION:
This study will evaluate the clinical efficacy, safety and the performance of radiofrequency heating and ultrasound delivered by the BTL-585-2 applicator of the BTL-585F system for non-invasive treatment of facial wrinkles and correcting facial skin laxity. The study is a prospective multicenter single-blinded two-arm study. The subjects will be enrolled and assigned into two study groups; group A (RF & US) and B (only RF) which will receive a treatment with different settings. Subjects of both groups will be required to complete four (4) treatment visits and two to three follow-up visits.

At the baseline visit, health status will be assessed and, if needed, additional tests will be performed. Inclusion and exclusion criteria will be verified and informed consent will be signed. Skin hydration and elasticity in the treatment area will be measured. In addition photographs of the treated area will be taken.

The treatment administration phase in both study groups will consist of four (4) treatment visits, delivered 7 - 14 days apart. Group A will receive treatment with active ultrasound (ON) and the intensity of radiofrequency will be set to a maximum tolerable level. The group B will receive treatment with the intensity of radiofrequency set to a maximum tolerable level, but without active ultrasound (OFF).

At every treatment visit after the first, prior to the procedure, the participants will be assessed for adverse effects resulting from the previous treatment(s) with the BTL-585F device.

At the last therapy visit, photographs of the treated area will be taken. In addition, subjects will receive Subject Satisfaction Questionnaire and Therapy Comfort Questionnaire to fill in. Skin hydration and elasticity in the treatment area will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects over 21 years of age seeking treatment and reduction of facial wrinkles and facial skin laxity
* Subjects should be able to understand the investigative nature of the treatment, the possible benefits and side effects, and must sign the Informed Consent Form
* Presence of clearly visible wrinkles in the treated area when the face is relaxed as deemed appropriate by the Investigator
* Subjects willing and able to abstain from partaking in any facial treatments other than the study procedure during study participation
* Willingness to comply with study instructions, to return to the clinic for the required visits, and to have photographs of their face taken

Exclusion Criteria:

* Bacterial or viral infection, acute inflammations
* Impaired immune system
* Isotretinoin in the past 12 months
* Skin related autoimmune diseases
* Radiation therapy and/or chemotherapy
* Poor healing and unhealed wounds in the treatment area
* Metal implants
* Permanent implant in the treated area
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
* Facial dermabrasion, facial resurfacing, or deep chemical peeling in the treatment area within 6 months prior to the treatment
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* History of any type of cancer
* Active collagen diseases
* Cardiovascular diseases (such as vascular diseases, peripheral arterial disease, thrombophlebitis and thrombosis)
* Pregnancy/nursing or IVF procedure
* History of bleeding coagulopathies, use of anticoagulants
* Any active condition in the treatment area, such as sores, psoriasis, eczema, rash and rosacea
* Any surgical procedure in the treatment area within the last three months or before complete healing
* Poorly controlled endocrine disorders, such as diabetes
* Acute neuralgia and neuropathy
* Kidney or liver failure
* Sensitivity disorders in the treatment area
* Varicose veins, pronounced edemas
* Prior use of dermal fillers, botulinum toxin, lasers, etc. therapies in the treated area that can influence the study results at the investigator discretion
* Unwillingness/inability to not change their usual cosmetics and especially not to use ani-aging or anti-wrinkles products in the treated area during the duration of the study including the follow-up period
* Any other disease or condition (e.g. eye disease) at the investigator discretion that may pose risk to the patient or compromise the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Overall Wrinkle Severity Change assessed according to the Fitzpatrick Wrinkle and Elastosis Scale (FWES) up to 3 months posttreatment follow-up | 3 months
  The Fitzpatrick Wrinkle and Elastosis Scale is a clinically validated assessment tool and will be used to assess skin wrinkle severity and elastosis on a scale from 1 to 9 (minimum 1 and maximum 9), where the lower score is considered better.
Change in overall facial appearance assessed according to the Global Aesthetic Improvement Scale (GAIS) up to 3 months posttreatment follow-up | 3 months
  Three independent evaluators will evaluate before and after photographs and grade them for change. Using the same photographs, they will evaluate changes in overall facial appearance according to the Global Aesthetic Improvement scale.
  For reporting of outcomes, the higher the GAIS value, the greater the improvement in the range -1 to 3.
  The following criteria will be used:
  Grade 3: Very Much Improved Grade 2: Much Improved Grade 1: Improved Grade 0: No Change Grade -1: Worse.

SECONDARY OUTCOMES:
Assessment of the safety profile by recording adverse events and assessing the subject's discomfort and pain | 3 months
  Occurrence of adverse events and side effects will be observed. Subjects experiencing a treatment-related adverse event (AE) in the first 90 days post-treatment, incidence/rates described as a percentage of the subjects.
Assessment of therapy comfort after the final study treatment based on a Therapy Comfort Questionnaire | up to 8 weeks
  A 5-point Likert scale Therapy Comfort Questionnaire and a numerical analog scale (NAS) will be used for evaluating comfort during the treatment sessions. The answers to the questions related to the subjects' overall skin and facial appearance will vary from "strongly agree (5)" to "strongly disagree (1)". The Therapy Comfort Questionnaire will be given to subjects at the final therapy visit.
Assessment of subject's satisfaction with study treatment using the Subject Satisfaction Questionnaire | 3 months
  A 5-point Likert scale Subject Satisfaction Questionnaire will be used to evaluate the participant's satisfaction with the therapy outcome. The answers to the questions related to the subjects' overall skin and facial appearance will vary from "strongly agree (5)" to "strongly disagree (1)". Subject satisfaction will be assessed after the last therapy visit and during the 1-month and 3-month follow-up visits.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - BOYD Beauty, Birmingham, Michigan
  - Refresh Dermatology, Houston, Texas

IPD SHARING:
Plan to Share IPD: No